CLINICAL TRIAL: NCT03546504
Title: Program to Improve Dental Care in Children With ASD: Reducing Sensory Stimulation and Building Oral Hygiene Habits
Brief Title: Program to Improve Dental Care: Children With ASD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: ran out of money
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lorie Richards, Chair and Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_0085018
Record Dates: First submitted 2018-05-14; First posted 2018-06-06 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Autism
Keywords: child; dental; oral health; sensory desensitization; sensory processing; occupational therapy
MeSH Terms: conditions — Autistic Disorder | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Single group pre-post-follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dental procedures modification and OT (Experimental): Modifying dental environment and procedures to reduce sensory stimulation. Occupational therapy provides desensitization techniques around the dental visit and home oral hygiene and habit training for oral hygiene activities.
  Interventions: Behavioral: Procedure alteration and occupational therapy

INTERVENTIONS:
Behavioral: Procedure alteration and occupational therapy — Modification of the dental environment and procedures to decrease sensory stimulation. Occupational therapy (8 weeks; 2x/week): sensory desensitization, habit training, social stories around dental visits

SUMMARY:
Children, aged 5-12, with autism spectrum disorder (ASD) who have difficulty with dental visits and daily oral hygiene will complete 3 dental assessments at baseline, 3 months, and 6 months. The dental environment and dental procedures will be altered based on the work of Cermak. In between the baseline and 3 months appointments, they will receive 8 weeks of occupational therapy targeting desensitization around dental activities and oral hygiene training. Post testing will assess the number of caries and overall oral health, the number of dental activities able to be accomplished without sedation, and the change in burden of caregivers to achieve oral hygiene.

DETAILED DESCRIPTION:
After providing consent and assent from applicable children, the researchers will administer the Sensory Processing Measure to test for sensory processing difficulties. Those that meet criteria on this assessment will then complete baseline testing. If the child does not score as having sensory processing problems on the Sensory Processing Measure, the family will be thanked for their time and withdrawn from the study. Their data will be destroyed and only that they were an interested family that failed screening due to lack of sensory processing problems recorded (no identifying information recorded). For those families that pass this screen, the caregivers will complete the following study measures Vineland Adaptive Behavior Scales, Dental Subscale of the Childrens Fear Survey, the Sensory Profile, the Screen for Child Anxiety Related Disorders, and study occupational therapists will complete an occupational performance evaluation (observing actual oral hygiene activities to assess skill level and determine barriers and supports for performance, interviewing parents for oral hygiene and dental visit history how they handle child's behavior that interferes with oral hygiene and dental visit activities, and gathering information about what rewards motivate the child using the Reinforcer Assessment for Individuals with Severe Disabilities. The oral hygiene activities observations serve as baseline data and information for clinical treatment planning, as well as research data. Information about parent reactions to child behaviors is clinical data that is necessary for individualizing occupational therapy treatment. The caregivers will be asked to videotape a typical oral hygiene session at home to be scored for the child's behavior by the researchers. The children will then complete a standard of care preventative dental visit (cleaning, X-rays, periodontal health check). The dental researcher will record the Decayed, Missing, Filled Surfaces (DMFS) Index, the Simplified Oral Hygiene Index, the Modified Gingival index from the Community Periodontal Index, and the child will be administered the Wong-Baker Faces Scale to measure discomfort. The dentist will obtain a saliva sample to test for bacteria associated with caries risk. The sample will be collected by having the child spit or drool into a cup. The saliva is analyzed on-site using a kit. That session will be videotaped for later scoring of behaviors. The dental research staff will fill out the Frankl Behavioral Scale describing the dental visit. The children will be scheduled for 8 sensory-based occupational therapy sessions, once per week, over 10 weeks. These sessions will be geared towards developing skills to discriminate, modulate, and integrate input from their multiple sensory systems, adapting their home environment and oral hygiene tasks to provide greater structure and reducing noxious sensory stimulation, and practicing of oral hygiene tasks using behavior learning techniques. By increasing their ability to properly interpret sensory input, we are increasing their ability to adapt to and respond to stimuli (self-regulation). Examples of activities that may be used include: increased input to muscles and joints through yoga or other weight bearing activities; oral desensitization for those that may have adverse responses (often specific textures); teaching coping techniques to decrease anxiety when presented with perceived adverse stimuli. The caregiver will be given a home program consisting of a sensory activity schedule everyday at home. These activities are specifically chosen and placed into a program to provide input to the sensory system that will help self-regulation. Activities can include: wall push-ups to provide increased input to the muscles and joints; utilizing a vibrating toothbrush to decrease oral sensitivity; warm baths; smelling specific scents. A visual schedule will be given to parents to use during tooth brushing at home to aid the participant in completing the task. These are typical occupational therapy services for children with life skill difficulties due to sensory processing problems. At the last session, occupational therapy research staff will complete study questionnaires. The occupational therapy sessions will primarily take place at the Division of Occupational Therapy's Life Skills Clinic, but up to 2 sessions may occur at the child's home if the occupational therapist deems that providing the therapy in the home would offer greater benefit to the child than all the session taking place at the clinic. After the 8 sessions of occupational therapy, the caregiver will be asked to videotape another typical oral hygiene session at home within 2 weeks of final occupational therapy session.

Then, the child will return to the dentist office for a 2nd preventative dental visit within 1 month at which the level of plaque, gingivitis, caries, fear, and cooperativeness with the dental procedures will be assessed. Two weeks before the follow-up dental appointment, parents will be sent a social story, about what to expect from the dental visit, to read with their child twice per day. At the 2nd dental visit, the teeth will be cleaned as well as assessed, but no X-rays will be taken. At this visit the dental environment and procedures will be modified to provide a better amount and type of sensory stimulation to the child. Examples may include the use of a weighted apron for deep proprioceptive input, which can be calming, using a head lamp rather than the typical dental light, providing headphones with soothing sounds playing, etc. This visit will be videotaped and dental research staff and caregivers will fill out study questionnaires as they did at baseline. The occupational therapist will also re-evaluate the child on the study outcome measures, observe the child tooth brushing and flossing, and interview the parent with the formal questionnaires and semi-structured interview.

Six months later, the child will have a 3rd preventative dental visit (with modifications as described above), which will be videotaped and with dental staff and caregivers filling out study questionnaires. The teeth will be assessed and cleaned, but no x-rays taken consistent with standard care procedures of x-rays only 1x/year. All dental visits will occur at the pediatric dental clinic at the Noorda Oral Health Sciences building. At the 6 month dental visit, parents will again be interviewed for changes in the ease of completing and quality of daily hygiene routines and perceived changes in tolerance for preventative dental visits and OT will again perform study outcome measures and observations with the child and caregiver.

If any dental caries are found during this period, they will be taken care of per standard of care dental procedures. If a child is found to need major restorative dental procedures during this study, he or she will be withdrawn from the study (although still offered standard clinical care) as the noxious sensation associated with a lot of dental procedures would confound the results of this study.

ELIGIBILITY:
Inclusion Criteria:

1. aged 5-12
2. able to follow 1-step verbal directions
3. able to reliably answer simple yes/no questions
4. have sensory processing difficulties as indicated by atypical scores on the Sensory Processing Measure [ref]
5. has difficulty completing oral hygiene and dental visits
6. has sufficient motor skills to brush own teeth
7. family is fluent in English
8. has a caregiver willing to adhere to home program

7) caregiver is willing to bring child to clinic 8 weekly occupational therapy clinic sessions

Exclusion Criteria:

1. unable to communicate
2. unable to physically handle toothbrush to brush teeth
3. requires extensive restorative dental work or has had such work within the past 3 months
4. has braces, temporary orthodontic prosthesis (e.g., retainers)
5. Greater than mild uncorrected hearing or visual impairments
6. uncontrolled seizures
7. has additional other neurodevelopmental conditions other than ADHD and Anxiety

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Child's behavior in typical oral hygiene activities | 1 month post-intervention
  digital recordings of children during oral hygiene activities coded within 10 second intervals for on-task behavior, aggression, agitation, time to complete activity - more on-task behavior, less aggression, less agitation, duration of activity closer to 5-10 minutes represents better functioning
Decayed, Missing, Filled Surfaces (DMFS) Index | 6 months post-intervention
  record of caries and missing teeth from dental exam; higher number means poorer oral health
Simplified Oral Hygiene Index | 1 month post-intervention
  dental report of oral health - Scored on a 0-3 scale with 0 = no debris and 3 = soft debris over > 2/3 of tooth; lower scores represent better oral health
Modified Gingival index from the Community Periodontal Index | 1 month post-intervention
  report of level of gingivitis - scored on a 0-4 scale with 0 = normal, no inflammation and 4 = severe inflammation; lower scores represent better oral health
Assessment of saliva for bacteria content | 1 month post-intervention
  collection of drool and bacterial assay - greater the bacteria count, the worse the oral health status
Number of dental procedures completed | 1 month post-intervention
  count of the number of dental procedures completed without sedation - greater the number of typical procedures, the better the functioning

SECONDARY OUTCOMES:
Dental Subscale of the Childrens Fear Survey | 1 month post-intervention
  rating by parent of child's fear associated with dental visits; 15 items are scored by selecting the "not afraid at all", " a little afraid", "a fair amount afraid", "pretty much afraid", or "very afraid"; lower amounts of fear represent better functioning
Frankl Behavioral Scale | 1 month post-intervention
  measures dentist perception of child's behavior during the dental visit: scored by rating child's behavior at this visit on 1-4 scale with 1= definitely negative and 4 = definitely positive; higher score = better behavior
Child's behavior during dental visits | 1 month post-intervention
  recording and coding of child behavior during dental visits - refusals, aggression, agitation - fewer of these represents better functioning
Parent report of burden of oral hygiene activities | 1 month post-intervention
  interview with parent related to burden of assisting child complete oral hygiene activities - reports of less burden represent better functioning
Parent report of burden of oral hygiene activities | 6 months post-intervention
  interview with parent related to burden of assisting child complete oral hygiene activities - report of less burden represents better functioning
Wong-Baker Faces Scale | 1 month post-intervention
  ratings of pain - used to measure discomfort during dental visit - lower score means less pain and discomfort
Wong-Baker Faces Scale | 6 months post-intervention
  ratings of pain - used to measure discomfort during dental visit - lower score means less pain and discomfort
Child's behavior in typical oral hygiene activities | 6 months post-intervention
  digital recordings of children during oral hygiene activities coded within 10 second intervals for on-task behavior, aggression, agitation, time to complete activity - more on-task behavior, less aggression, less agitation, duration of activity closer to 5-10 minutes represents better functioning
Simplified Oral Hygiene Index | 6 months post-intervention
  dental report of oral health - Scored on a 0-3 scale with 0 = no debris and 3 = soft debris over > 2/3 of tooth; lower scores represent better oral health
Modified Gingival index from the Community Periodontal Index | 6 months post-intervention
  report of level of gingivitis - scored on a 0-4 scale with 0 = normal, no inflammation and 4 = severe inflammation; lower scores represent better oral health
Assessment of saliva for bacteria content | 6 months post-intervention
  collection of drool and bacterial assay - greater the bacteria count, the worse the oral health status
Dental Subscale of the Childrens Fear Survey | 6 months post-intervention
  rating by parent of child's fear associated with dental visits; 15 items are scored by selecting the "not afraid at all", " a little afraid", "a fair amount afraid", "pretty much afraid", or "very afraid"; lower amounts of fear represent better functioning
Frankl Behavioral Scale | 6 months post-intervention
  measures dentist perception of child's behavior during the dental visit: scored by rating child's behavior at this visit on 1-4 scale with 1= definitely negative and 4 = definitely positive; higher score = better behavior
Child's behavior during dental visits | 6 months post-intervention
  recording and coding of child behavior during dental visits - refusals, aggression, agitation - fewer of these represents better functioning
Number of dental procedures completed | 6 months post-intervention
  greater the number of typical procedures, the better the functioning

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cermak SA, Stein Duker LI, Williams ME, Dawson ME, Lane CJ, Polido JC. Sensory Adapted Dental Environments to Enhance Oral Care for Children with Autism Spectrum Disorders: A Randomized Controlled Pilot Study. J Autism Dev Disord. 2015 Sep;45(9):2876-88. doi: 10.1007/s10803-015-2450-5. PMID 25931290
- [Result] Duker LIS, Henwood BF, Bluthenthal RN, Juhlin E, Polido JC, Cermak SA. Parents' perceptions of dental care challenges in male children with autism spectrum disorder: An initial qualitative exploration. Res Autism Spectr Disord. 2017 Jul;39:63-72. doi: 10.1016/j.rasd.2017.03.002. Epub 2017 May 20. PMID 29098015